CLINICAL TRIAL: NCT04141878
Title: Dementia and Diabetes Prevention Program (DDPP)
Brief Title: Dementia and Diabetes Prevention Program
Acronym: DDPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: East Oakland Sports Center (Unknown); Tice Creek Fitness Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1464339
Record Dates: First submitted 2019-10-15; First posted 2019-10-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Dementia
Keywords: Diabetes; Dementia; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Dementia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either the Aerobic Exercise Group or the Diet Skills Group. Each participant will eventually complete both groups.
Masking Description: There is no masking in this study. Everyone will know whether the participant is currently participating in the Aerobic Exercise Group or the Diet Skills Group. All participants will eventually complete both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Active Comparator): Participants will follow a structured program that includes exercise 3 times per week for about 30 minutes each time. The type of aerobic exercise will vary, but will primarily focus on in-class walking tutorials. Participants will work with a Personal Trainer to create their own physical activity program that will fit their needs and schedule. The Personal Trainer will supervise the participants directly for the first 6 weeks. Once participants are consistently and safely meeting their goals, their Personal Trainer will allow unsupervised exercise sessions.
  Interventions: Behavioral: Aerobic Exercise
- Diet Skills Group (Active Comparator): Participants will attend weekly classes focused on incorporating heart healthy foods (e.g., fruits and vegetables) into their existing dietary plan. We will ask them to limit the number of calories they take in and will show them how to use portion control with the goal of losing body weight. Participants will also learn hands-on skills for preparing healthy meals at home in cooking classes led by professional chefs.
  Interventions: Behavioral: Diet Skills

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants will follow a structured program that includes exercise 3 times per week for about 30 minutes each time. The type of aerobic exercise may vary, but will primarily focus on walking tutorials.
  Arms: Aerobic Exercise Group
Behavioral: Diet Skills — Participants will attend weekly classes focused on incorporating heart healthy foods into their existing diets. Calories will be restricted, and portion control will be taught with the goal of losing body weight. Hands-on skills will be taught for preparing healthy home-cooked meals by professional chefs.
  Arms: Diet Skills Group

SUMMARY:
This is a multicenter, randomized 2-arm clinical trial of two lifestyle interventions varying in intensity and format, in 400 older African American and non-Hispanic whites at increased risk of cognitive decline and dementia in the East San Francisco Bay Area. The trial will include two lifestyle interventions that differ in intensity and format:

1. Aerobic Exercise (AEx) Intervention that involves aerobic activities with in-class walking workouts and tutorials and carried out at the East Oakland Sports Center (EOSC) and Tice Creek Fitness Center (TICE).
2. Dietary counseling to support adherence to the Mediterranean-Diet Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) diet to encourage increased consumption of berries, green leafy and other vegetables, whole grains, nuts, fish, poultry, beans and olive oil, and to reduce consumption of fried/fast foods, red meat, whole fat cheese, sweets, butter and trans-fat margarines.

DETAILED DESCRIPTION:
The 8-month diet and AEx regimens used here are theoretically motivated by implementation science and use the best available practices to treat multisystemic disabling processes. The recent Centers for Disease Control (CDC) review of Diabetes Prevention Program (DPP) implementation literature found that 1 hour per week is the optimal length and frequency to balance cost and attentional demands of the participants. DPP class structure generally involves a 10-min weigh-in, a discussion of adherence to personal weight loss and exercise goals, formal DPP content delivery, and lastly a discussion of barriers to adherence. Diet module content focuses on calorie restriction by altering the composition of participants' meals. These goals include reducing trans-fats, saturated fats, sodium, and carbohydrates and increasing fruits, vegetables, whole grains, and fiber. Participants set weight reduction goals for themselves with personalized goals between 5% and 10% of total body weight dependent on the participant's level of obesity - effectively replacing prepared foods with traditional (Mediterranean) diet.

Because cognitive abilities do not appear to change without a corresponding improvement in cardio respiratory (CR) fitness, the 8-month AEx module content optimizes CR fitness improvement with in-class walking workouts and tutorials. All health instructors at TICE and EOSC will have at least an Associates level degree in exercise physiology and be required to have personal training certification. They will always be under the direct supervision of the PI. Direct supervision of the participants by these health instructors will occur for all exercise sessions until the weekly duration target of 150 minutes a week is reached (Week 6). We introduce more flexibility in scheduling exercise when the participant is consistently and safely meeting their goals by allowing unsupervised exercise sessions at the facility when exercise trainers may not be available (i.e. early morning, nights, and weekends). Participants are still required to have at least one directly supervised exercise session per week to maintain contact with program staff and encourage adherence to the program. Unsupervised exercise sessions are conducted similarly to supervised exercise and session data will be reviewed by the exercise instructor at the weekly supervised session.

Per a well-developed literature on DPP best practices,159,160 we will limit intervention class sizes to about 20 people. Over the course of 5 years, we will run 30 to 35 full DPP groups, each session meeting weekly for 20 consecutive weeks of diet-focused or AEx-focused intervention.

Previous studies suggest that salivary hormones such as cortisol, alpha-amylase and testosterone all measure glucocorticoid (GC) sensitivity, a potent biomarker of age-related stress. We will measure three stress markers in spit before and after a participant exercises during the 6-minute walk challenge at baseline and at each follow-up visit. Because better fitness is believed to improve one's reaction to stressful events, changes in these hormones may reflect the adaptation of a person's ability to cope with emotional and physical stress as they become more cardiorespiratory fit.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (as per the Telephone Assessment of Physical Activity)
* Poor diet (as per the MIND Diet Screener)
* Cognitive function: absence of significant cognitive impairment as per the modified Telephone Interview for Cognitive Status (TICSm; age-, education-, and race-adjusted TICSm >32)
* Lives in a region where the DDPP interventions will be delivered
* Does not plan to travel outside of the home geographic area for more than 3 months over the course of the study
* Free of physical disabilities that preclude participation in the study
* Willing to complete all study-related activities for 32 weeks
* Willing to be randomized to either lifestyle intervention group

Exclusion Criteria:

* Age <60
* Body Mass Index (BMI) >40
* Any significant neurologic disease, including any form of dementia, Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma with persistent neurologic sequelae or known structural brain abnormalities
* History of major depression within the last 12 months
* History of bipolar disorder or schizophrenia as per Diagnostic and Statistical Manual of Mental Disorders (DSM) V criteria
* History of alcohol or substance abuse or dependence within the past 2 years, as per DSM V criteria
* Use of psychoactive medications within the last 3 months including tricyclic antidepressants, antipsychotics, mood-stabilizing psychotropic agents (e.g., lithium salts), psychostimulants, opiate analgesics, antiparkinsonian medications, anticonvulsant medications (except gabapentin and pregabalin for non-seizure indications), systemic corticosteroids, or medications with significant central anticholinergic activity; in the absence of major depression, stable dose use of selective serotonin reuptake inhibitors or serotonin and norepinephrine reuptake inhibitors are allowed
* Health profiles that would jeopardize their safety to participate: (Screen failures will be referred immediately to a physician for medical examination): (1) Myocardial infarction or symptoms of unstable coronary artery disease (e.g., angina) in the last six months, (2) Uncontrolled hypertension within the past 6 months, (3) Morbid obesity (BMI<40), (4) History of clinically-evident stroke, (5) Clinically-significant infection within the past 30 days, (6) Significant pain or musculoskeletal disorder limiting the ability to participate safely, or (7) Clinically significant
* Past or current use of insulin to treat type 2 diabetes
* Serious diabetic event within 6 months of enrollment
* Lung disease requiring either regular use of corticosteroids or the use of supplemental oxygen (inhaled steroids for asthma is permissible)
* Renal disease
* Clinically significant abnormalities in laboratory blood tests as per judgment of the Study Physician
* History within the last 2 years of treatment for primary or recurrent malignant disease, excluding non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment
* History of hip fracture, joint replacement, or spinal surgery in the last 6 months
* Currently receiving physical therapy or cardiopulmonary rehabilitation
* History of a malabsorptive bariatric procedure (gastric bypass, biliopancreatic diversion); other bariatric procedures involving restriction (i.e., sleeve, band) are not exclusionary
* For women: currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months
* Currently incarcerated
* Receiving hospice care
* Adults unable to provide consent for participation
* PI/Study Physician discretion regarding appropriateness of participation or concern about intervention adherence

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Change in DDPP Neuropsychological Test Battery | Change from Baseline to Month 4
  Cognitive Performance

SECONDARY OUTCOMES:
Change in 6-Minute Walk Test | Change from Baseline to Month 4
  A reliable estimate of cardiorespiratory fitness that measures the maximum distance a person can walk in 6 minutes and the change in heart rate from start to finish.
Change in Hand-Grip Strength | Change from Baseline to Month 4
  Grip strength is determined using a hand-held dynamometer and measured in kilograms (kg) of isometric force. Participants are then required to squeeze the hand-held dynamometer inner and outer grips towards each other as hard as possible without bending the elbow, while remaining seated.
Change in Chair Rise | Change from Baseline to Month 4
  Measure of lower body strength. Participants are seated in a chair without armrests and instructed to rise from the chair to a stand and sit down again. The process is repeated as many times as possible for 30 seconds.
Change in Body Mass Index (BMI) | Change from Baseline to Month 4
  weight, height, and waist circumference measurements are collected and BMI calculated.
Change in Glycated Hemoglobin (Hemoglobin A1C) | Change from Baseline to Month 4
  hemoglobin A1C will be analyzed using the University of California, Davis (UCD) Alzheimer's Disease Center (ADC) site Finger stick whole blood analyzer

CONTACTS AND LOCATIONS:
Overall Officials: David K Johnson, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Alzheimer's Disease Center, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers.

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/dementia-diabetes-prevention-program-ddpp-940291/